CLINICAL TRIAL: NCT03488069
Title: Sedation Practices and Preferences of Turkish Intensive Care Physicians: National Survey
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, seval urkmez, Principal Investigator, Istanbul University
Other Study IDs: 261075
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness; Sedation
Keywords: critical care; sedation; practice; survey
MeSH Terms: conditions — Critical Illness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Submission of survey answers

SUMMARY:
Sedation is one of the most common practices applied in intensive care units (ICU) and the management of sedation, analgesia and delirium is a quality measure in ICUs. Several intensive care societies published guidelines regarding the use of sedatives and analgesics recently. In literature there are many survey studies investigating practices of sedation in ICUs of different countries, but knowledge of the sedation practices of intensive care physicians in Turkey is lacking. The aim of this study was to provide a baseline knowledge on this matter and to establish some points to be improved. An electronic survey form, consisting of 34 questions was generated with google forms, posted to 1700 email addresses and 429 returned (25%). The survey included questions about demographics and choices and routines of sedation, analgesia, neuromuscular blockers and delirium administration. Ninety-six percent of the respondents indicated that they practiced sedation in their ICUs and mechanical ventilation was checked as the primary indication (94%). On the question regarding drug choices for sedation, midazolam was the most preferred agent (90%). About pain questions, the most used evaluation tool was visual analogue scale (69.0%) and 83% of the respondents preferred to use tramadol for pain, followed by paracetamol (81.6%). Of the participants, 50.5% indicated that they routinely evaluated delirium and 56% of them used confussion assessment method for ICU. The awareness of 2013 American College of Critical Care Medicine (ACCM) guideline for the management of pain, agitation, and delirium was only 38%. The results of this survey have indicated some areas to be improved, such as low incidence of written sedation protocols, frequent use of benzodiazepines, and delirium screening. A national guideline should be prepared taking pain, agitation, and delirium in focus.

DETAILED DESCRIPTION:
This national survey study and questionnaire was approved by the institutional ethics committee of Istanbul University, Cerrahpasa Medical School (approval nr. 261075, date 07.07.2017).

An electronic survey form consisting of 34 questions was generated with google forms (https://docs.google.com/forms) after a literature search with search words "sedation" and "practice" and "survey".

The first part of the form included questions about demographics, intensive care, and hospital characteristics. The second part contained questions on choices and routines of sedation administration, which multiple choices could be indicated.

The questions were first pilot tested for misunderstandings with the ICU physicians in two intensive care units, and the link for the survey was posted to all email addresses registered in the Turkish Society of Intensive Care member database (1700 members) on 2.8.2017. A second notification was sent to same email addresses on 16.10.2017 with a notice of not to reply the survey if it was replied after the first email. Participation in the survey was voluntary and anonymous, and there was no compensation for participation.

Accepting responses to the survey was stopped in 01/11/2017, and answers were downloaded from the web site.

Statistical Analysis The answers were analyzed using Excel spreadsheets (Microsoft Corporation, Redmond, WA, USA). The demographic data are expressed as mean (±SD) and counts and percentages. The answers regarding sedation practices are expressed as counts and percentages. No statistical comparisons had been made as this was a descriptive study.

ELIGIBILITY:
Inclusion Criteria:

* All physicians accepting to participate the survey

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All intensive care physicians that are the member of Turkish Society of Intensive Care
Sampling Method: Non-Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Practices and preferences of sedation | 3 months
  Collection of answers to the survey

CONTACTS AND LOCATIONS:
Overall Officials: seval urkmez, MD, Principal Investigator — IU, Cerrahpasa Medical School, Dept of Intensive Care
Locations (1):
- Istanbul University Cerrahpasa Medical School, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Urkmez S, Erdogan E, Utku T, Dikmen Y. Sedation Practices and Preferences of Turkish Intensive Care Physicians: A National Survey. Turk J Anaesthesiol Reanim. 2019 Jun;47(3):220-227. doi: 10.5152/TJAR.2019.49799. Epub 2019 Feb 24. PMID 31183469